CLINICAL TRIAL: NCT05011721
Title: Digital Phenotyping (Physical Activity, Heart Rate, Sleep) in Young Breast Cancer Patients Treated With Neoadjuvant Chemotherapy
Brief Title: Digital Phenotyping in Young Breast Cancer Patients Treated With Neoadjuvant Chemotherapy
Acronym: NeoFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2020-20
Record Dates: First submitted 2021-07-19; First posted 2021-08-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: neoadjuvant; digital; prevention; activity tracker
MeSH Terms: conditions — Breast Neoplasms | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with activity tracker (Experimental): Women allocated to the intervention arm will used an activity tracker
  Interventions: Device: Activity tracker

INTERVENTIONS:
Device: Activity tracker — Participants will receive a Withings Steel HR activity tracker (Withings, Issy-les-Moulineaux, France), which they will be asked to wear 24 hours per day throughout the whole intervention (12 months). At baseline, the Withings Health Mate mobile phone application will be downloaded onto each participant's smartphone or tablet. The clinical research assistant will instruct the participant in the use of the activity tracker. The participant will then accept and activate the sharing of the data collected with the secure server dedicated to the "NeoFit" study at the Institut Curie. Participants will be asked to synchronize the activity tracker regularly (ideally daily) via Bluetooth with the Withings Health Mate application, for automatic transfer of the data to the secure "NeoFit" space.

SUMMARY:
NeoFit is a prospective, national, multicenter, single-arm open-label study. It will include a total of 300 participants under the age of 70 years treated with neoadjuvant chemotherapy for BC. Participants will receive a Withing Steel HR activity tracker, which they will be asked to wear 24 h per day for 12 months. The principal assessments will be performed at baseline, at the end of neoadjuvant chemotherapy and at 12 months. The investigators will evaluate clinical (e.g. toxicity, efficacy of chemotherapy), lifestyle, quality of life, fatigue, and physical activity parameters. All questionnaires will be completed on a REDCap form, via a secure internet link.

DETAILED DESCRIPTION:
BACKGROUND: In young women, breast cancer (BC) has particular characteristics, such as a more advanced stage at diagnosis, aggressive tumor characteristics, and a poorer prognosis. NeoFit aims to use an activity tracker to identify and describe various digital profiles (physical activity, heart rate, sleep) in women under 70 years of age treated with neoadjuvant chemotherapy for BC.

METHODS: NeoFit is a prospective, national, multicenter, single-arm open-label study. It will include a total of 300 participants under the age of 70 years treated with neoadjuvant chemotherapy for BC. Participants will receive a Withing Steel HR activity tracker, which they will be asked to wear 24 h per day for 12 months. The principal assessments will be performed at baseline, at the end of neoadjuvant chemotherapy and at 12 months. The investigators will evaluate clinical (e.g. toxicity, efficacy of chemotherapy), lifestyle, quality of life, fatigue, and physical activity parameters. All questionnaires will be completed on a REDCap form, via a secure internet link.

DISCUSSION: NeoFit will make it possible, through the use of an activity tracker, to visualize changes, over a one-year period, in the lifestyle of young women treated for BC by neoadjuvant chemotherapy. This exploratory study will provide fundamental knowledge about the digital phenotypes of young BC patients treated with NAC and their relationships to chemotherapy toxicity and efficacy. This trial will pave the way for interventional studies on physical activity and sleep interventions.

ELIGIBILITY:
Inclusion criteria :

* female
* ≥ 18 years old and <70 years old
* histologically confirmed BC, whatever the histological subtype (hormone receptor positive (RH+), negative (RH-), with (HER2+) overexpression or without (HER2-) HER2 overexpression, or triple negative)
* planned NAC (up to the day of the first neoadjuvant chemotherapy treatment)
* Eastern Cooperative Oncology Group Performance status ≤2
* willing to participate for the entire duration of the study
* ability to use a compatible smartphone or Tablet PC to download the application Withings Health Mate (from iOS 10 and Android 5.0 or above)
* Internet access
* valid health insurance
* able to read, write and understand French

Exclusion criteria :

* presence of metastases
* Presence of bilateral breast cancer
* a history of cancer other than basal cell skin lesions and cervical dysplasia
* pregnancy, likelihood of pregnancy, or breastfeeding
* impossibility of follow-up throughout the study for medical, social, family, geographic or psychological reasons
* deprived of liberty through a judicial or administrative decision.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Describe physical activity profiles in breast cancer patients under 70 years of age treated by neoadjuvant chemotherapy | Month 12
  The activity tracker will register step counts for each day. the investigators will plot the average daily step counts and the 95% confidence interval across the entire study period. Then will will study the change in step count trajectory during the study. Linear mixed model will be used for describing change over time
Describe heart rate profiles in breast cancer patients under 70 years of age treated by neoadjuvant chemotherapy | Month 12
  The activity tracker will register heart rate at 10-minute intervals for each day. The investigators will plot the average heart rate frequency and the 95% confidence interval across the entire study period. Then will will study the change in heart rate frequency trajectory during the study. Linear mixed model will be used for describing change over time
Describe sleep profiles in breast cancer patients under 70 years of age treated by neoadjuvant chemotherapy | Month 12
  The activity tracker will register sleep duration for each day. The investigators will plot the average sleep duration and the 95% confidence interval across the entire study period. Then will tudy the change in sleep duration trajectory during the study. Linear mixed model will be used for describing change over time
Identify digital profiles (physical activity, heart rate, sleep) in breast cancer patients under 70 years of age treated by neoadjuvant chemotherapy | Month 12
  To identify digital profiles, The investigators will combine step counts profiles, heart frequency profiles and sleep profiles using mixed models with latent classes. The use of a mixed model will make it possible to analyze repeat data for the population, and to determine an average profile or trajectory for the whole population. The optimal number of classes will be determined a posteriori, based on a set of statistical and clinical criteria. The most widely used statistical criterion is the "Bayesian information criterion" (BIC), which penalizes the model's likelihood according to its complexity. The BIC, which is stricter than many other criteria, has been shown to have a better performance in simulations. The number of trajectories will also be based on clinical interpretation (whether it is worthwhile retaining classes containing very small numbers of subjects, etc.).

SECONDARY OUTCOMES:
Analyze the effects of digital profiles on treatment toxicity | End of neoadjuvant chemotherapy, Month 12
  Occurence of severe toxicity (grade >2) according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) Tests will be performed to compare means (Student's t test), or categorical variables (chi2test). The investigators will also perform multinomial logistic regression analyses with univariate and multivariate models, to determine the probability of belonging to a class relative to the corresponding reference class
Analyze the effects of digital profiles on quality of life | End of neoadjuvant chemotherapy, Month 12
  Quality of life will be assessed with the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) Quality of Life Questionnaire (EORTC QLQ-C30) version 3 validated in 2000, a multidimensional questionnaire validated for use with cancer patients. The QLQC30 questionnaire contains 30 items assessing five functional domains (physical, role, emotional, cognitive, and social), one overall quality-of-life domain, three symptom domains (pain, fatigue and nausea), and six individual items (dyspnea, insomnia, anorexia, diarrhea, constipation, and financial impact). Participants will respond on a Likert scale ranging from "not at all" to "very much" and from "very poor" to "excellent" for the overall quality-of-life questions only. Scores will be standardized on a scale of 0 to 100, according to the EORTC scoring manual. Higher scores correspond to better functioning, a better overall quality of life and more symptoms.
Analyze the effects of digital profiles on fatigue | End of neoadjuvant chemotherapy, Month 12
  The multidimensional aspects of fatigue will be evaluated with the EORTC QLQ-FA12 version 1 module, which was validated for cancer-related fatigue in 2017. EORTC QLQ-FA12 contains 12 items assessing the physical, cognitive, and emotional domains of cancer-related fatigue. Participants will complete a four-point Likert-scale questionnaire, with responses ranging from "not at all" to "very much". All scores will be transformed to a scale of 0 to 100, with higher scores indicating a greater degree of fatigue. The estimated completion time for this questionnaire is five minutes.
  Tests will be performed to compare means (Student's t test), or categorical variables (chi2test). The investigators will also perform multinomial logistic regression analyses with univariate and multivariate models, to determine the probability of belonging to a class relative to the corresponding reference class
Develop models for predicting toxicity during the course of treatment | End of the neoadjuvant chemotherapy, Month 12
  The prediction of treatment toxicity will be assessed by CTCAE v4.0.
Develop models for predicting fatigue changes during the course of treatment | End of the neoadjuvant chemotherapy, Month 12
  The prediction of fatigue will be assessed by change from baseline in fatigue scores on FA12 questionnaire and at the end of the neoadjuvant chemotherapy and at 12 months..
Develop models for predicting quality of life changes during the course of treatment | End of the neoadjuvant chemotherapy, Month 12
  The prediction of a deterioration of the quality of life will be assessed by change in the global score in EORTC QLQC30 questionnaire from baseline and at the end of the neoadjuvant chemotherapy and at 12 months..

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Reyal, MD, Principal Investigator — Institut Curie
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Background] Delrieu L, Hamy AS, Coussy F, Kassara A, Asselain B, Antero J, De Villele P, Dumas E, Forstmann N, Guerin J, Hotton J, Jouannaud C, Milder M, Leopold A, Sedeaud A, Soibinet P, Toussaint JF, Vercamer V, Laas E, Reyal F. Digital phenotyping in young breast cancer patients treated with neoadjuvant chemotherapy (the NeoFit Trial): protocol for a national, multicenter single-arm trial. BMC Cancer. 2022 May 4;22(1):493. doi: 10.1186/s12885-022-09608-y. PMID 35509030